CLINICAL TRIAL: NCT05080049
Title: Erythropoietin to Improve Critical Care Patient Outcomes: Feasibility Study of a Multicenter, Randomized, Placebo-controlled Trial of Subcutaneous Erythropoietin Injection for Intensive Care Patients
Brief Title: Erythropoietin to Improve Critical Care Patient Outcomes
Acronym: EPO-ICU-FS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPO-ICU-FS
Record Dates: First submitted 2021-09-20; First posted 2021-10-15 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Anemia; Intensive Care
Keywords: Anemia; Intensive Care; Feasibility study; Erythropoietin
MeSH Terms: conditions — Anemia | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erythropoietin (Experimental): Erythropoietin alpha or theta 40,000 UI (1 ml) sc each week if Hb <12 g/dL (for maximum 5 weeks)
  Interventions: Drug: Erythropoietin
- Placebo (Placebo Comparator): saline sc injection (1 ml) each weeks if Hb <12 g/dL, for a maximum of 5 weeks,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin — Patients receive a subcutaneous injection of 40,000 IU of erythropoietin alfa or zêta, repeated weekly until Day 28 (if the hemoglobin level is <12 g/dl and the patient remains hospitalized).
  The study treatments are administered by an open-label nurse. In both groups, before each injection, iron deficiency (defined as reticulocyte Hb <29 pg, or hepcidin <41 µg/L, or ferritin <100 µg/L, or ferritin <300 µg/L with transferrin saturation <20%) is treated with intravenous iron infusion (depending on the product available at the center). A restrictive transfusion strategy is recommended as long as the patient remains in the ICU, according to recent recommendations.
  Six visits are scheduled: V1 for inclusion and the first injection, V2 at Day 7(±2 days) for the second injection, V3 at Day 14(±2 days) for the third injection, V4 at Day 21(±2 days) for the fourth injection, V5 at Day 28(±2 days) for the fifth injection.
  Arms: erythropoietin
Drug: Placebo — In the control arm, patients receive a subcutaneous injection of placebo (0.9% NaCl) according to the same schedule.
  The study treatments are administered by an open-label nurse. In both groups, before each injection, iron deficiency (defined as reticulocyte Hb <29 pg, or hepcidin <41 µg/L, or ferritin <100 µg/L, or ferritin <300 µg/L with transferrin saturation <20%) is treated with intravenous iron infusion (depending on the product available at the center). A restrictive transfusion strategy is recommended as long as the patient remains in the ICU, according to recent recommendations.
  Six visits are scheduled: V1 for inclusion and the first injection, V2 at Day 7(±2 days) for the second injection, V3 at Day 14(±2 days) for the third injection, V4 at Day 21(±2 days) for the fourth injection, V5 at Day 28(±2 days) for the fifth injection.
  Arms: Placebo

SUMMARY:
Recently, the french societies for critical care (SFAR and SRLF) produced guidelines for anemia treatment in critically ill patients that recommend the use of erythropoietin (EPO) in these patients, but the european society (ESICM) recommended against the use of EPO in this patients, despite recent meta analysis showing a lower mortality in patients treated with EPO.

Nevertheless, RCT on EPO in the ICU are quite all, new data are thus needed. Before conducting a large study on EPO in anemic patients in the ICU, we propose to cinduct a feasability RCT to evaluate the feasability of such a study.

DETAILED DESCRIPTION:
Anemia is very common in intensive care patients, affecting approximately two-thirds of patients on admission, with a mean admission hemoglobin (Hb) level of 11.0 g/dl. The severity of anemia is associated with increased morbidity and mortality. Its pathophysiology is complex, involving blood loss (from repeated blood sampling, invasive procedures, surgical interventions, etc.) and inflammation. The latter is responsible for a decrease in endogenous erythropoietin (EPO) production and a decreased bone marrow response, which can be very prolonged (half of the patients discharged from ICU with anemia are still anemic at 6 months of discharge, with low levels of EPO, compared to the observed Hb levels). On this basis, several randomized clinical trials (RCTs) evaluating the effect of EPO on the transfusion rate in this population were performed in the 1990s-2000s. The authors showed a modest reduction in blood transfusion, which was not considered clinically relevant in view of the cost of EPO at that time.

Since then, meta-analyses evaluating the benefits and risks of EPO in intensive care patients suggest a positive impact of EPO on mortality. The largest, including 34 studies (and 930,470 patients) reports a reduction in the relative risk of mortality of 0.76, 95% CI [0.61 - 0.92]. Beyond the reduction in red blood cell transfusions, the benefit of EPO could be directly due to its erythropoietic effect (correction of anemia) and/or its anti-inflammatory/anti-apoptotic properties. Based on this literature, the French critical care societies have recently recommended the use of EPO. However, the European Society of Intensive Care Medicine (ESICM) recently recommended against the use of EPO, based on the same literature, but suggested that the benefit of EPO should be evaluated. Indeed, the main obstacle to recommending the use of EPO seems to be economic, whereas the arrival on the market of biosimilar molecules has significantly reduced these costs.

Most of the trials on EPO in critical care patients (and included in the meta-analyses) are quite old (about 15 years) and none of them had mortality as primary endpoint. In addition, transfusion practices and the quality of blood products have changed significantly over the years. In this context of disagreement on the recommendations for the use of EPO in these patients, but of potential benefit on mortality, there is an urgent need to evaluate whether EPO decreases mortality in adult anemic patients admitted to intensive care. However, calculation of the number of patients needed to evaluate the benefit of EPO on mortality in this population yields a number of patients to be included of the order of 1800-2000 patients.

Before considering the implementation of a multicenter study involving such a large number of patients, a pilot study evaluating the feasibility and inclusion capacity for such a study seems indispensable according to the latest CONSORT recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years),
* admitted to intensive care for more than 72 hours and less than 7 days
* who have received invasive ventilatory support and/or treatment with a vasoactive agent for at least one day since admission
* with an Hb level < 12 g/dl,
* with consent from the patient or patient's relative (or emergency inclusion procedure).

Exclusion Criteria:

* Moribund patient,
* Current hospitalization for acute coronary syndrome,
* Recent history of thromboembolic event (< 3 months),
* Uncontrolled hypertension despite adequate antihypertensive therapy,
* Myelodysplasia or chronic pathology requiring iterative transfusions,
* EPO treatment within the last 30 days,
* Participation in another interventional trial of an erythropoiesis-stimulating agent or anemia treatment,
* Expected discharge from the intensive care unit within 24 hours,
* Known hypersensitivity to EPO or any of its components,
* A history of erythroblastopenia following erythropoietin therapy
* Pregnant, breast-feeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person under a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 90 days
  ≥50% of eligible patients will need to be enrolled, but the trial will not be feasible if the inclusion rate is ≤ 25% or less
Adherence to allocation groups | 90 days
  A high level of matching of randomization and group allocation should be achieved, with at least 85% of included patients receiving protocol-allocated treatment, but if ≤ 65% patients receive protocol-allocated treatment, the trial is not feasible
Completion of follow-up of included patients | 90 days
  ≥ 85% of patients should be followed through to the end of follow-up, but if <65% patients are followed through to the last visit, the protocol will not be feasible

SECONDARY OUTCOMES:
The proportion of patients lost to follow-up at each visit | 7, 14, 21, 28 and 90 days
  The proportion of patients lost to follow-up at each visit
The rate of missing data for mortality outcome | 90 days
  The rate of missing data for mortality outcome
The rate of compliance with the therapeutic protocol at each visit for inpatients | 7, 14, 21, and 28 days
  The rate of compliance with the therapeutic protocol at each visit for inpatients
Mean serum hemoglobin value | 28 days
  Mean serum hemoglobin value
ICU mortality | up to 90 days
  ICU mortality
Hospital mortality | up to 90 days
  Hospital mortality
ICU length of stay | up to 90 days
  ICU length of stay
Hospital length of stay | up to 90 days
  Hospital length of stay
Blood transfusion | 90 days
  Proportion of patients who received at least one red blood cell transfusion
number of red blood cells transfused | 90 days
  number of red blood cells transfused
90 days survival analysis | 90 days
  90 days survival analysis
Occurrence of hospital readmission (censored at 90 days after inclusion), | 90 days
  at least one hospital readmission after the hospital discharge
Number of days living at home (or previous place of living) | 90 days
  Number of days living at home (or previous place of living) at D90
Quality of life measured by the EQ-5D 5L scale, EuroQol 5 dimensions | 90 days
  The value from this scale records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine'. The scale is rated from 0 to 100.
Proportion of patients with a thromboembolic event | 90 days
  Thrombolic event: pulmonary embolism, venous or arterial thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Léger, MD, Principal Investigator — Angers University Hospital; Sigismond Lasocki, MD, Study Director — Angers University Hospital
Locations (2):
- France (2):
  - Cholet Hospital, Cholet
  - UH Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided
Yes